CLINICAL TRIAL: NCT01517555
Title: A Single Centre, Randomised, Double-blind, Placebo Controlled Trial to Evaluate the Possible Drug-drug Interaction Between Liraglutide and Paracetamol and the Effects of Liraglutide on Postprandial Glucose and Insulin, Gastric Emptying, Appetite Sensations and Energy Intake in Subjects With Type 2 Diabetes
Brief Title: Effect of Liraglutide on Absorption of Paracetamol in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN2211-1698; 2006-000561-10 (EudraCT Number)
Record Dates: First submitted 2012-01-21; First posted 2012-01-25 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Liraglutide; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Liraglutide (Experimental)
  Interventions: Drug: liraglutide; Drug: placebo; Drug: paracetamol
- Placebo (Placebo Comparator)
  Interventions: Drug: liraglutide; Drug: placebo; Drug: paracetamol

INTERVENTIONS:
Drug: liraglutide — Administered as a subcutaneous injection. Initial dose 0.6 mg daily, adjusted to 1.2 mg daily in week 2 and escalated to 1.8 mg daily in week 3
Drug: placebo — Administered as a subcutaneous injection. Given as daily volume of 100 mcl, 200 mcl and 300 mcl respectively
Drug: paracetamol — One single dose of 1 g. Tablet

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to to investigate if there is a drug-drug interaction between liraglutide and paracetamol (Benuron®) and to investigate the effect of liraglutide on post prandial glucose.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus
* Diet-treated subjects with type 2 diabetes with HbA1c 7.5-9.5 %
* Subjects with type 2 diabetes in oral anti-diabetic drug (OAD) monotherapy treated with metformin or alpha-glucosidase inhibitors with HbA1c 7.0-9.5%
* Body mass index (BMI) 18.5-40 kg/m^2
* Subjects should have a stable body weight for at least 3 months prior to screening (as judged by the Investigator)

Exclusion Criteria:

* Impaired liver function
* Impaired renal function
* Clinically significant active cardiovascular disease including history of myocardial infarction within the last 6 months and/or heart failure
* Any clinically significant abnormal ECG (electrocardiogram)
* Uncontrolled treated/untreated hypertension
* Recurrent severe hypoglycaemia as judged by the Investigator
* Active hepatitis B and/or active hepatitis C
* Positive human immunodeficiency virus (HIV) antibodies
* Known or suspected allergy to trial product(s) or related products

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2006-10; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Area under the curve of paracetamol
Area under the curve of post prandial plasma glucose

SECONDARY OUTCOMES:
Area under the curve of paracetamol
Cmax, maximum concentration
tmax, time to reach Cmax
t½, terminal half-life
Terminal elimination rate constant
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Neuss, Germany

REFERENCES:
- [Result] Kapitza C, Zdravkovic M, Hindsberger C, Flint A. The effect of the once-daily human glucagon-like peptide 1 analog liraglutide on the pharmacokinetics of acetaminophen. Adv Ther. 2011 Aug;28(8):650-60. doi: 10.1007/s12325-011-0044-y. Epub 2011 Jul 20. PMID 21792552
- [Result] Flint A, Kapitza C, Hindsberger C, Zdravkovic M. The once-daily human glucagon-like peptide-1 (GLP-1) analog liraglutide improves postprandial glucose levels in type 2 diabetes patients. Adv Ther. 2011 Mar;28(3):213-26. doi: 10.1007/s12325-010-0110-x. Epub 2011 Feb 17. PMID 21340616
- [Result] Flint A, Kapitza C, Zdravkovic M. The once-daily human GLP-1 analogue liraglutide impacts appetite and energy intake in patients with type 2 diabetes after short-term treatment. Diabetes Obes Metab. 2013 Oct;15(10):958-62. doi: 10.1111/dom.12108. Epub 2013 Apr 23. PMID 23551925
- [Result] Roge RM, Klim S, Ingwersen SH, Kjellsson MC, Kristensen NR. The Effects of a GLP-1 Analog on Glucose Homeostasis in Type 2 Diabetes Mellitus Quantified by an Integrated Glucose Insulin Model. CPT Pharmacometrics Syst Pharmacol. 2015 Jan;4(1):e00011. doi: 10.1002/psp4.11. Epub 2014 Dec 30. PMID 26225223
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com